CLINICAL TRIAL: NCT01257841
Title: Effects of Four-day Fast on Gut-derived Hormones and Inflammatory Markers in Healthy, Normal-weight Women.
Brief Title: Secondary Analysis of Gut Hormones and Inflammatory Cytokines in Fasting Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Steven K Grinspoon, M.D. Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2002P-000518SA1
Record Dates: First submitted 2010-12-07; First posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Fasting; Gut hormones; Inflammatory Cytokines
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fasting alone (Placebo Comparator)
  Interventions: Behavioral: Fasting
- Fasting plus leptin (Active Comparator)
  Interventions: Drug: Leptin administration; Behavioral: Fasting

INTERVENTIONS:
Drug: Leptin administration — Leptin 0.05 mg/kg sc daily in divided doses (0800, 1400, 2000, and 0200h) for four days.
  Arms: Fasting plus leptin
Behavioral: Fasting — Complete fasting, save for water and multivitamin, for four days.

SUMMARY:
The original study executed between 2002-2004 was an interventional trial in which 20, healthy, normal-weight female subjects were randomized to a four-day fast plus daily subcutaneous injections of leptin or a four day fast plus daily subcutaneous injections of a placebo. The primary endpoints were gonadotropin pulsatility, TSH secretion and thyroid function, and cortisol secretion. The current study is a secondary analysis focussed on the placebo group which underwent a four-day fast. The study is looking at the effects of fasting on gut-derived hormones and inflammatory markers in healthy, normal-weight women. The hypothesis for this secondary analysis was that four days of fasting would augment levels of orexigenic gut-derived hormones and suppress levels of anorexigenic gut-derived horomones, while suppressing secretion of inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* female age 18-35
* BMI 20-26.0
* eumenorrheic with normal FSH, TSH, Prolactin
* Hgb > 12 g/dL, normal creatinine
* normal puberty and development
* negative pregnancy test. In addition, subjects agreed not to be sexually active during the course of the inpatient study and to use contraception for a period of 48 hours after discharge from the hospital.

Exclusion Criteria:

* medical or endocrine problems known to affect thyroid, reproductive, GH or cortisol function
* medications known to affect neuroendocrine function
* prior history of eating disorder or significant menstrual irregularities
* subjects who have a known hypersensitivity to E. Coli derived protein.
* subjects with a history of seizure disorder, significant cardiac disease, medication for cardiac disease, or kidney disease
* history of anaphylaxis or anaphylactoid like reactions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Hormone levels change from baseline. | Change from baseline after 4 days of intervention.
  Original study looking at gonadotropin pulsitility, TSH secretion and thyroid function, and cortisol secretion. Present study looking at gut-hormone secretion.

SECONDARY OUTCOMES:
Levels of inflammatory cytokines change from baseline. | Change from baseline after 4 days of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts

REFERENCES:
- [Result] Canavan B, Salem RO, Schurgin S, Koutkia P, Lipinska I, Laposata M, Grinspoon S. Effects of physiological leptin administration on markers of inflammation, platelet activation, and platelet aggregation during caloric deprivation. J Clin Endocrinol Metab. 2005 Oct;90(10):5779-85. doi: 10.1210/jc.2005-0780. Epub 2005 Aug 2. PMID 16076944
- [Result] Schurgin S, Canavan B, Koutkia P, Depaoli AM, Grinspoon S. Endocrine and metabolic effects of physiologic r-metHuLeptin administration during acute caloric deprivation in normal-weight women. J Clin Endocrinol Metab. 2004 Nov;89(11):5402-9. doi: 10.1210/jc.2004-1102. PMID 15531489
- [Result] Koutkia P, Schurgin S, Berry J, Breu J, Lee BS, Klibanski A, Grinspoon S. Reciprocal changes in endogenous ghrelin and growth hormone during fasting in healthy women. Am J Physiol Endocrinol Metab. 2005 Nov;289(5):E814-22. doi: 10.1152/ajpendo.00093.2005. Epub 2005 Jun 21. PMID 15972272